CLINICAL TRIAL: NCT05909904
Title: A Randomized, Phase 2, Open-Label, Multi-Arm Study of Tislelizumab in Combination With Investigational Agents as First-Line Treatment in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of Tislelizumab in Combination With Investigational Agents in Participants With Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-HNSCC-201; CTR20232123 (Other: ChinaDrugTrials); 2023-503418-63-00 (EU CTIS Number)
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tislelizumab (Active Comparator): Tislelizumab 200 milligrams (mg) administered once every 3 weeks
  Interventions: Drug: Tislelizumab
- Tislelizumab + BGB-A425 (Experimental): Tislelizumab 200 mg administered once every 3 weeks with BGB-A425
  Interventions: Drug: Tislelizumab; Drug: BGB-A425
- Tislelizumab + LBL-007 (Experimental): Tislelizumab 200 mg administered once every 3 weeks with LBL-007
  Interventions: Drug: Tislelizumab; Drug: LBL-007
- Tislelizumab + BGB-A425 + LBL-007 (Experimental): Tislelizumab 200 mg administered once every 3 weeks with BGB-A425 and LBL-007
  Interventions: Drug: Tislelizumab; Drug: BGB-A425; Drug: LBL-007

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously
  Other Names: BGB-A317
Drug: BGB-A425 — Administered intravenously
  Other Names: Surzebiclimab
  Arms: Tislelizumab + BGB-A425; Tislelizumab + BGB-A425 + LBL-007
Drug: LBL-007 — Administered intravenously
  Other Names: Alcestobart
  Arms: Tislelizumab + BGB-A425 + LBL-007; Tislelizumab + LBL-007

SUMMARY:
This study is designed to evaluate the efficacy and safety of tislelizumab and tislelizumab in combination with investigational agent(s) in first-line recurrent or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
This study will test whether tislelizumab alone and combined with other investigational agents can be used to improve treatment outcomes in participants with head and neck squamous cell carcinoma. The main goals of the study are to determine how many participants may no longer have evidence of cancer or have some improvement in the signs and symptoms of cancer after treatment and to determine what adverse events, or side effects, participants might experience.

Tislelizumab is used to block the programmed cell death protein-1 pathway so that immune system cells (T-cells) can better protect the body from infection and find tumor cells to attack. Tislelizumab may be used in combination with other therapies as a promising approach with potential therapeutic benefits to treat participants with cancer. The study will enroll approximately 160 participants. Participants will be randomly assigned (by chance, similar to flipping a coin) to one of the various treatment groups. Tislelizumab and investigational agents will be administered as an infusion through a vein at regularly scheduled intervals.

The study will take place at multiple centers worldwide. Treatments will continue until participants experience no benefits, too many side effects, or withdraw consent.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed R/M HNSCC that is considered incurable by local therapies

  1. The eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx
  2. Participants should not have had prior systemic therapy administered in the R/M setting; systemic therapy which was completed prior to randomization/enrollment if given as part of multimodal treatment for locally or locoregionally advanced disease is allowed
* Participants must have positive PD-L1 expression (Combined Positive Score [CPS] ≥ 1)
* Have at least 1 measurable lesion as defined per RECIST v1.1
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Adequate hematologic and organ function as indicated by specific laboratory values within 7 days of first dose of study drug
* Willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of study drug(s)

Exclusion Criteria:

* Recurrent or metastatic carcinoma of the nasopharynx (any histology), squamous cell carcinoma of unknown primary, squamous cell carcinoma that originated from the skin and salivary gland primary tumor or non-squamous histologies (eg, mucosal melanoma)
* Prior therapy with an anti-PD-1, anti-PD-L1, PD-L2, T-cell immunoglobulin and TIM-3, LAG-3, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
* Any active malignancy ≤ 2 years before randomization/enrollment except for the specific cancer under investigation in this study, those with a negligible risk of metastasis or death, and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, localized prostate cancer, and carcinoma in situ of the cervix or breast)
* History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including pulmonary fibrosis, and acute lung diseases
* A history of severe hypersensitivity reactions to other monoclonal antibodies or has experienced a severe immune-mediated adverse event (imAE), an imAE that led to treatment discontinuation, or a cardiac or ocular imAE of any grade with prior immunotherapy

Note: Other inclusion and exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 3 years and 6 months
  ORR is defined as percentage of participants who have a confirmed complete response (CR) or a confirmed partial response (PR) as assessed by the investigators using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 3 years and 6 months
  PFS is defined as the time from the date of randomization to the date of the first documentation of progressive disease assessed by the investigators per RECIST v1.1 or death, whichever occurs first
Duration of Response (DOR) | Up to approximately 3 years and 6 months
  DOR is defined as the time from the first determination of a confirmed response per RECIST v1.1 until the first documentation of progression or death, whichever occurs first
Clinical Benefit Rate (CBR) | Up to approximately 3 years and 6 months
  CBR is defined as the percentage of participants with a best overall response of a confirmed CR, a confirmed PR, or a durable stable disease (SD) (SD duration ≥ 24 weeks)
Disease Control Rate (DCR) | Up to approximately 3 years and 6 months
  DCR is defined as the percentage of participants with a best overall response of a confirmed CR, a confirmed PR, or SD
Number of Participants with Adverse Events | Up to approximately 3 years and 6 months
  Number of participants with adverse events, including laboratory values, vital signs, physical examinations, and electrocardiogram findings
Overall Survival (OS) | Up to approximately 3 years and 6 months
  OS is defined as the time from the date of randomization to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (73):
- United States (9):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Stanford Medicine, Stanford, California
  - Rocky Mountain Cancer Centers, Llp(Us Oncology Research), Lone Tree, Colorado
  - Florida Cancer Specialist Research Institute Lake Nona, Orlando, Florida
  - Florida Cancer Specialist Research Institute Panhandle, Tallahassee, Florida
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Oncology and Hematology Associates of Southwest Virginia, Inc (Us Oncology Research), Blacksburg, Virginia
  - Cancer Care Northwest, Spokane Valley, Washington
  - Northwest Cancer Specialist, Pc(Us Oncology Research), Vancouver, Washington
- Australia (7):
  - Nepean Hospital, Kingswood, New South Wales
  - North Shore Private Hospital, St Leonards, New South Wales
  - Gold Coast Private Hospital, Gold Coast, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
  - Northeast Health Wangaratta, Wangaratta, Victoria
  - St John of God, Murdoch, Murdoch, Western Australia
- Canada (2):
  - British Columbia Cancer Agency the Vancouver Centre, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
- China (22):
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - Beijing Tongren Hospital, Cmu, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (4):
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Paris, Paris
  - Ico Site Rene Gauducheau, SaintHerblain
  - Institut Gustave Roussy, Villejuif
- Arensia Exploratory Medicine Llc, Tbilisi, Georgia
- Italy (4):
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Istituto Europeo Di Oncologia, Milan
  - Scientific Institute of Pavia Maugeri, Pavia
  - Istituto Clinico Humanitas, Rozzano
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (7):
  - Keimyung University Dongsan Hospital, Dalseogu, Daegu Gwang'yeogsi
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
- Spain (4):
  - Ico Lhospitalet Hospital Duran I Reynals, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Thailand (4):
  - Ramathibodi Hospital Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
  - Songklanagarind Hospital (Prince of Songkhla University), Hat Yai
  - Srinagarind Hospital (Khon Kaen University), Muang
- Turkey (Türkiye) (2):
  - Tr Trakya University Health Research and Application Center (Hospital), Edirne
  - Medical Park Izmir Hospital, Izmir
- United Kingdom (2):
  - Royal Marsden Hospital, London
  - Royal Marsden Hospital Sutton, Sutton